CLINICAL TRIAL: NCT02280044
Title: Double Blind, Placebo-Controlled Trial Assessing the Efficacy of Rifaximin in Preventing Campylobacteriosis in Subjects Challenged With Campylobacter Jejuni
Brief Title: Efficacy of Rifaximin in Preventing Campylobacteriosis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: Naval Medical Research Center (U.S. Federal Agency); Uniformed Services University of the Health Sciences (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CIR296
Record Dates: First submitted 2014-10-29; First posted 2014-10-31 (Estimated); Results first posted 2018-11-20 (Actual); Last update posted 2018-11-20 (Actual); Status verified 2018-10

CONDITIONS: Dysentery; Diarrhea; Enteric Campylobacteriosis
Keywords: Campylobacter jejuni; rifaximin; antibiotic prophylaxis; dysentery; diarrhea
MeSH Terms: conditions — Dysentery; Diarrhea; Campylobacter Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- rifaximin (Experimental): Subjects receiving rifaximin prophylaxis will be challenged with C. jejuni
  Interventions: Biological: Rifaximin intervention
- placebo (Placebo Comparator): Subjects receiving placebo will be challenged with C. jejuni
  Interventions: Biological: Placebo intervention

INTERVENTIONS:
Biological: Rifaximin intervention — Rifaximin administered then Challenge with C jejuni
  Arms: rifaximin
Biological: Placebo intervention — Placebo administered then Challenge with C jejuni
  Arms: placebo

SUMMARY:
This study is a randomized, double-blinded, placebo-controlled, in-patient trial evaluating the prophylactic efficacy of rifaximin against campylobacteriosis following challenge with C. jejuni.

DETAILED DESCRIPTION:
30 healthy volunteers (2 of these were planned alternates) gave informed consent and were enrolled to participate in a study to determine the efficacy of prophylactic rifaximin in preventing diarrheal illness following challenge with C. jejuni, strain CG8421. Volunteers were screened for inclusion and exclusion criteria and were admitted to the inpatient unit of the Center for Immunization Research at Johns Hopkins University. Volunteers were treated with rifaximin or placebo in a double blind manner for four days, beginning the day prior to challenge. On the day of challenge, the volunteers were given 5x10(5) C. jejuni with bicarbonate buffer and were then monitored and treated for any symptoms. Stools were cultured daily for the excretion of C. jejuni and all subjects were treated with antibiotics to insure that the challenge strain has cleared prior to to discharge. Subjects were followed for six months following the inpatient phase to detect adverse events following the study.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female between 18 and 50 years of age, inclusive
2. General good health, without significant medical illness, abnormal physical examination findings or clinically significant laboratory abnormalities, as determined by the PI (may consult with the Research Monitor on a case-by-case basis)
3. Demonstrate comprehension of the protocol procedures and knowledge of Campylobacter illness by passing a written examination (pass grade ≥ 70%)
4. Willing to participate after informed consent obtained
5. Available for all planned follow-up visits and remain available for clinic visits (for examination, blood draws and stool collection) and monitoring for 90 days post-challenge and by phone for 180 days post-challenge
6. If the subject is female, she is eligible to enter if she is of:

   * Non-childbearing potential (i.e., physiologically incapable of becoming pregnant, including any female who is post-menopausal. For purposes of this study, postmenopausal is defined as one year without menses); or must have documentation of having undergone tubal ligation or hysterectomy. OR
   * Childbearing potential; has a negative serum pregnancy test at screening and a negative urine pregnancy test on admission (Study Day -1), and agrees to the use of an efficacious hormonal or barrier method of birth control during the study, abstinence is acceptable

Exclusion Criteria:

General health/issues

1. Presence of a significant medical condition (e.g., psychiatric conditions; gastrointestinal disease, such as peptic ulcer,symptoms or evidence of active gastritis/dyspepsia, inflammatory bowel disease, irritable bowel syndrome (as defined by the Rome III criteria or medical diagnosis); alcohol or illicit drug abuse/dependency) or laboratory abnormalities which in the opinion of the investigator preclude participation in the study
2. Evidence of Immunoglobulin A deficiency (serum IgA < 7 mg/dL or below the limit of detection of assay)
3. Positive serology results for HIV, HBsAg, or Hepatitis C virus antibodies
4. Positive urine toxicology screen
5. Significant abnormalities in screening laboratory hematology or serum chemistry, as determined by PI or PI in consultation with the Research Monitor and sponsor
6. Use of any medication known to affect the immune function (e.g., corticosteroids and others) within 30 days preceding receipt of the challenge inoculum or planned to be used during the active study period
7. Nursing mother on the day of admittance to the inpatient unit

Study-specific exclusionary conditions based on potential increased risk or complicating outcome ascertainment. (See protocol details for complete list of exclusions.)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2014-10; Primary Completion 2016-08-09 (Actual); Study Completion 2016-08-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kawsar Talaat, M.D., Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Center for Immunization Research, Johns Hopkins Bloomberg School of Public Heatlh, Baltimore, Maryland, United States

REFERENCES:
- [Result] Kirkpatrick BD, Lyon CE, Porter CK, Maue AC, Guerry P, Pierce KK, Carmolli MP, Riddle MS, Larsson CJ, Hawk D, Dill EA, Fingar A, Poly F, Fimlaid KA, Hoq F, Tribble DR. Lack of homologous protection against Campylobacter jejuni CG8421 in a human challenge model. Clin Infect Dis. 2013 Oct;57(8):1106-13. doi: 10.1093/cid/cit454. Epub 2013 Jul 9. PMID 23840001
- [Result] Riddle MS, Gutierrez RL, Verdu EF, Porter CK. The chronic gastrointestinal consequences associated with campylobacter. Curr Gastroenterol Rep. 2012 Oct;14(5):395-405. doi: 10.1007/s11894-012-0278-0. PMID 22864805
- [Result] Tribble DR, Baqar S, Scott DA, Oplinger ML, Trespalacios F, Rollins D, Walker RI, Clements JD, Walz S, Gibbs P, Burg EF 3rd, Moran AP, Applebee L, Bourgeois AL. Assessment of the duration of protection in Campylobacter jejuni experimental infection in humans. Infect Immun. 2010 Apr;78(4):1750-9. doi: 10.1128/IAI.01021-09. Epub 2010 Jan 19. PMID 20086085
- [Result] Tribble DR, Baqar S, Carmolli MP, Porter C, Pierce KK, Sadigh K, Guerry P, Larsson CJ, Rockabrand D, Ventone CH, Poly F, Lyon CE, Dakdouk S, Fingar A, Gilliland T, Daunais P, Jones E, Rymarchyk S, Huston C, Darsley M, Kirkpatrick BD. Campylobacter jejuni strain CG8421: a refined model for the study of Campylobacteriosis and evaluation of Campylobacter vaccines in human subjects. Clin Infect Dis. 2009 Nov 15;49(10):1512-9. doi: 10.1086/644622. PMID 19842970
- [Result] Poly F, Read TD, Chen YH, Monteiro MA, Serichantalergs O, Pootong P, Bodhidatta L, Mason CJ, Rockabrand D, Baqar S, Porter CK, Tribble D, Darsley M, Guerry P. Characterization of two Campylobacter jejuni strains for use in volunteer experimental-infection studies. Infect Immun. 2008 Dec;76(12):5655-67. doi: 10.1128/IAI.00780-08. Epub 2008 Sep 22. PMID 18809665
- [Result] Flores J, Dupont HL, Jiang ZD, Okhuysen PC, Melendez-Romero JH, Gonzalez-Estrada A, Carrillo I, Paredes M. A randomized, double-blind, pilot study of rifaximin 550 mg versus placebo in the prevention of travelers' diarrhea in Mexico during the dry season. J Travel Med. 2011 Sep-Oct;18(5):333-6. doi: 10.1111/j.1708-8305.2011.00549.x. Epub 2011 Aug 1. PMID 21896097
- [Result] Martinez-Sandoval F, Ericsson CD, Jiang ZD, Okhuysen PC, Romero JH, Hernandez N, Forbes WP, Shaw A, Bortey E, DuPont HL. Prevention of travelers' diarrhea with rifaximin in US travelers to Mexico. J Travel Med. 2010 Mar-Apr;17(2):111-7. doi: 10.1111/j.1708-8305.2009.00385.x. PMID 20412178
- [Result] Steffen R, Sack DA, Riopel L, Jiang ZD, Sturchler M, Ericsson CD, Lowe B, Waiyaki P, White M, DuPont HL. Therapy of travelers' diarrhea with rifaximin on various continents. Am J Gastroenterol. 2003 May;98(5):1073-8. doi: 10.1111/j.1572-0241.2003.07283.x. PMID 12809830
- [Result] Infante RM, Ericsson CD, Jiang ZD, Ke S, Steffen R, Riopel L, Sack DA, DuPont HL. Enteroaggregative Escherichia coli diarrhea in travelers: response to rifaximin therapy. Clin Gastroenterol Hepatol. 2004 Feb;2(2):135-8. doi: 10.1016/s1542-3565(03)00322-7. PMID 15017618
- [Result] Armstrong AW, Ulukan S, Weiner M, Mostafa M, Shaheen H, Nakhla I, Tribble DR, Riddle MS. A randomized, double-blind, placebo-controlled study evaluating the efficacy and safety of rifaximin for the prevention of travelers' diarrhea in US military personnel deployed to Incirlik Air Base, Incirlik, Turkey. J Travel Med. 2010 Nov-Dec;17(6):392-4. doi: 10.1111/j.1708-8305.2010.00462.x. PMID 21050319
- [Result] Dupont HL, Jiang ZD, Belkind-Gerson J, Okhuysen PC, Ericsson CD, Ke S, Huang DB, Dupont MW, Adachi JA, De La Cabada FJ, Taylor DN, Jaini S, Martinez Sandoval F. Treatment of travelers' diarrhea: randomized trial comparing rifaximin, rifaximin plus loperamide, and loperamide alone. Clin Gastroenterol Hepatol. 2007 Apr;5(4):451-6. doi: 10.1016/j.cgh.2007.02.004. Epub 2007 Mar 26. PMID 17382603
- [Result] DuPont HL, Jiang ZD, Ericsson CD, Adachi JA, Mathewson JJ, DuPont MW, Palazzini E, Riopel LM, Ashley D, Martinez-Sandoval F. Rifaximin versus ciprofloxacin for the treatment of traveler's diarrhea: a randomized, double-blind clinical trial. Clin Infect Dis. 2001 Dec 1;33(11):1807-15. doi: 10.1086/323814. Epub 2001 Oct 23. PMID 11692292
- [Derived] Rimmer JE, Harro C, Sack DA, Talaat KR, Gutierrez RL, DeNearing B, Brubaker J, Laird RM, Poly F, Maue AC, Jaep K, Alcala A, Mochalova Y, Gariepy CL, Chakraborty S, Guerry P, Tribble DR, Porter CK, Riddle MS. Rifaximin Fails to Prevent Campylobacteriosis in the Human Challenge Model: A Randomized, Double-Blind, Placebo-Controlled Trial. Clin Infect Dis. 2018 Apr 17;66(9):1435-1441. doi: 10.1093/cid/cix1014. PMID 29145631

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Per protocol, a total of thirty subjects were admitted to the inpatient unit and randomized to receive investigational product on day -1 to ensure the target sample size was obtained. Two subjects received three doses of product but were discharged on Day 0 prior to challenge. Both subjects were randomized to the placebo arm.
Period: Overall Study
Arm/Group | Rifaximin | Placebo
Started | 15 | 15
Completed | 15 | 13
Not Completed | 0 | 2
Not completed — Planned alternate | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rifaximin | Placebo | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 30 [29 to 37] | 31 [26 to 41] | 31 [29 to 38]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 9
  Male | 11 | 10 | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  Race: American Indian or Alaska Native | 0 | 0 | 0
  Race: Asian | 0 | 0 | 0
  Race: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Race: Black or African American | 13 | 14 | 27
  Race: White | 1 | 1 | 2
  Race: More than one race | 1 | 0 | 1
  Race: Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Campylobacteriosis
Description: A clinical illness meeting at least one of the following patterns:
  * Moderate to severe diarrhea.
  * Fever (present on at least 2 occasions, at least 20 minutes apart) without diarrhea, plus an associated symptom (nausea, vomiting, abdominal cramps, tenesmus, or gross blood in ≥ 2 stools); with consideration of potential alternative diagnosis per clinical investigator based on illness time course and associated symptoms.
Time Frame: 120 hours after challenge
Measure: Count of Participants; unit: Participants
Arm/Group | Rifaximin | Placebo
Number analyzed (Participants) | 15 | 13
Participants | 13 | 11

2. Post Hoc Outcome: Recrudescent Events
Description: Recovered C jejuni from fecal specimen on follow-up after an apparent cure
Time Frame: 84 Days
Measure: Count of Participants; unit: Participants
Arm/Group | Rifaximin | Placebo
Number analyzed (Participants) | 15 | 13
Participants | 2 | 3

ADVERSE EVENTS:
Time Frame: 84 days
Arm/Group | Rifaximin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/13
Other Adverse Events (participants affected / at risk) | 13/15 | 13/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rifaximin (N=15) | Placebo (N=13)
Nausea (Gastrointestinal disorders) | 6 (6) | 9 (9)
Abdominal Cramps (Gastrointestinal disorders) | 9 (9) | 9 (9)
Abdominal pain (Gastrointestinal disorders) | 7 (7) | 7 (7)
anorexia (Gastrointestinal disorders) | 9 (9) | 8 (8)
Bilateral knees and elbows itching (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Bloating (Gastrointestinal disorders) | 3 (3) | 7 (7)
Diarrhea (outpatient) (Gastrointestinal disorders) | 2 (2) | 3 (3)
Dysentery (Gastrointestinal disorders) | 4 (4) | 8 (8)
Erythematous maculopapular rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Gas (Gastrointestinal disorders) | 1 (1) | 3 (3)
Vaginal Yeast infection (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Abdominal tenderness (Gastrointestinal disorders) | 3 (3) | 4 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (5) | 4 (4)
Blurred vision in right eye (Eye disorders) | 1 (1) | 0 (0)
Body aches (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Bowel sounds (Gastrointestinal disorders) | 3 (3) | 2 (2)
Campylobacter infection of recrudescence (Gastrointestinal disorders) | 2 (2) | 3 (3)
Campylobacter infection of recrudescence 2 (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chills (Immune system disorders) | 10 (10) | 8 (8)
Fecal Urgency (Gastrointestinal disorders) | 0 (0) | 1 (1)
Fever (Immune system disorders) | 8 (8) | 6 (6)
Gastric bubbling (Gastrointestinal disorders) | 2 (2) | 1 (1)
Headache (General disorders) | 9 (9) | 9 (9)
Hypotension (Cardiac disorders) | 1 (1) | 1 (1)
Lightheadedness (General disorders) | 5 (5) | 5 (5)
Malaise (General disorders) | 10 (10) | 8 (8)
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 8 (8) | 5 (5)
Pain with Defecation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Skin warm to touch (Skin and subcutaneous tissue disorders) | 0 (0) | 1
Swollen tender left wrist (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 5 (5) | 4 (4)
Tenesmus (Gastrointestinal disorders) | 1 (1) | 2 (2)
Vomiting (Gastrointestinal disorders) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes